CLINICAL TRIAL: NCT03645577
Title: Phrenic Nerve Injury During Pulmonary Vein Isolation With the Second-generation Cryoballoon: Clinical, Procedural, and Anatomical Characteristics
Brief Title: Phrenic Nerve Injury During Pulmonary Vein Isolation With the Second-generation Cryoballoon.
Acronym: YETI-Registry
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Collaborators: Principal Investigator: Roland Richard Tilz, MD (Unknown)
Responsible Party: Principal Investigator, Christian-H. Heeger, MD, PI, University of Luebeck
Other Study IDs: 18-151A
Record Dates: First submitted 2018-07-26; First posted 2018-08-24 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Phrenic Nerve Palsy
Keywords: Pulmonary vein isolation; Phrenic nerve palsy; Paroxysmal atrial fibrillation; Persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the most frequent complication associated with cryoballoon PVI. The main hypothesis is to explore the incidence of phrenic nerve palsy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* Cryoballoon PVI
* Periprocedural phrenic lesion

Exclusion Criteria:

- Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a PVI by the second generation Cryoballoon.
Sampling Method: Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of phrenic nerve palsy | 06/2012 until 04/2018
  The overall incidence of phrenic nerve palsy during second and third Generation Cryoballoon based PVI will be evaluated.

SECONDARY OUTCOMES:
Predictors of phrenic nerve palsy | 06/2012 until 04/2018
  Predictors for transient and permanent phrenic nerve palsy will be evaluated. For this purpose baseline characteristics (e.g. age, sex, BMI, CHADS-VASc-Score) as well as periprocedural data (e.g. minimal cryoballoon temp., cryoballoon temp. after 30 seconds, time to isolation, PV diameter, use of doublestopp technique and draw back manouever) will be assesseda and predictors will be calculated using adequat statistical techniques.
Clinical course of phrenic nerve palsy | 06/2012 until 04/2018
  The clincial course of phrenic nerve palsy after second and third Generation Cryoballoon based PVI will be evaluated by follow-up appointments according to each centers standard of care. For this purpose follow-up data will be evaluated and the clinical course will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart Center Luebeck, Electrophysiology, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heeger CH, Popescu SS, Sohns C, Pott A, Metzner A, Inaba O, Straube F, Kuniss M, Aryana A, Miyazaki S, Cay S, Ehrlich JR, El-Battrawy I, Martinek M, Saguner AM, Tscholl V, Yalin K, Lyan E, Su W, Papiashvili G, Botros MSN, Gasperetti A, Proietti R, Wissner E, Scherr D, Kamioka M, Makimoto H, Urushida T, Aksu T, Chun JKR, Aytemir K, Jedrzejczyk-Patej E, Kuck KH, Dahme T, Steven D, Sommer P, Tilz RR. Impact of cryoballoon application abortion due to phrenic nerve injury on reconnection rates: a YETI subgroup analysis. Europace. 2023 Feb 16;25(2):374-381. doi: 10.1093/europace/euac212. PMID 36414239
- [Derived] Heeger CH, Sohns C, Pott A, Metzner A, Inaba O, Straube F, Kuniss M, Aryana A, Miyazaki S, Cay S, Ehrlich JR, El-Battrawy I, Martinek M, Saguner AM, Tscholl V, Yalin K, Lyan E, Su W, Papiashvili G, Botros MSN, Gasperetti A, Proietti R, Wissner E, Scherr D, Kamioka M, Makimoto H, Urushida T, Aksu T, Chun JKR, Aytemir K, Jedrzejczyk-Patej E, Kuck KH, Dahme T, Steven D, Sommer P, Richard Tilz R. Phrenic Nerve Injury During Cryoballoon-Based Pulmonary Vein Isolation: Results of the Worldwide YETI Registry. Circ Arrhythm Electrophysiol. 2022 Jan;15(1):e010516. doi: 10.1161/CIRCEP.121.010516. Epub 2021 Dec 28. PMID 34962134